CLINICAL TRIAL: NCT01302795
Title: A Phase II Multi Center Open Label Pilot Study To Assess a Potential Effect of an Anti-Il-1-Beta Antagonist in the Treatment of Pyoderma Gangrenosum
Brief Title: Canakinumab for Pyoderma Gangrenosum
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DER-USZ-AAN-008
Record Dates: First submitted 2011-02-17; First posted 2011-02-24 (Estimated); Last update posted 2016-09-27 (Estimated); Status verified 2016-09

CONDITIONS: Pyoderma Gangrenosum
Keywords: Interleukin 1 beta; Canakinumab; autoinflammatory syndrome
MeSH Terms: conditions — Pyoderma Gangrenosum | interventions — canakinumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Canakinumab (Experimental): Canakinumab s.c. 150-300mg Week 0, (2), 8
  Interventions: Drug: Canakinumab

INTERVENTIONS:
Drug: Canakinumab — Monoclonal antibody inhibiting interleukin 1 beta
  Other Names: Ilaris

SUMMARY:
This study is a prospective open label evaluation of Canakinumab (Ilaris) for treatment of subjects with pyoderma gangrenosum.

DETAILED DESCRIPTION:
At the start of the study (week 0), all patients will receive one subcutaneous injection of 150mg Canakinumab. Patients are then going to be examined at weeks 2, 4, 8, 12 and 16.

At 2 weeks, all patients are going to be evaluated for response by Physician's global assessment (PGA) of the target lesion. Patients with PGA 0-1 are not going to receive another injection at this timepoint, while patients with PGA 2-4 are going to receive another 150mg Canakinumab.

At 4 weeks, in case of PGA 4, patients are going to be offered a first or second line drug as an alternative therapy (corticosteroids, cyclosporin A or infliximab, dosage see below "Alternative therapy in case of missing response") and stay within the trial (due to the long half-life of canakinumab) until week 8.

At week 8, patients with PGA 0 receive another 150mg Canakinumab only, and patients with PGA 4 are not going to receive additional study drug, but are strongly encouraged to attend following medical visits for observation until the end of the study and/or switch to a first or second line drug as alternative therapy (see below). All other patients with PGA 1-3 receive the total accumulative dose of Canakinumab that they had received on week 0 and 2, namely 150 or 300mg.

The study duration for each individual is going to be 16 weeks. At week 8 and 16, safety laboratory investigations with blood differential (Neutrophil granulocytes, monocytes, eosinophils, basophils, lymphocytes, thrombocytes, erythrocytes, hemoglobin), AST, ALT, y-GT, AP, Bilirubin (total), Creatinine, Na, K, CRP are going to be determined.

ELIGIBILITY:
Inclusion criteria: Patients fulfilling all of the following inclusion criteria may be enrolled in the study

1. Age = 18 years of age at visit 0 and
2. Subjects are capable of giving informed consent
3. Non-healing ulcer with primarily neutrophil infiltration, regardless of size and location
4. Diagnosis of pyoderma gangrenosum as confirmed by clinical and histological examination (see exclusion criteria). In case of doubt, a steering committee consisting of experts of the participating centers is going to evaluate whether inclusion is possible or not

Exclusion criteria:

* Other etiologies of ulcers 15, namely venous insufficiency, arterial occlusion, microcirculatory disorders, physical or chemical injury, infection, neuropathy, vasculitis, haematological disorders, neoplasia, other ulcerating diseases: Diseases with cutaneous manifestations mimicking pyoderma gangrenosum, including but not limited to Wegener's granulomatosis, polyarteritis nodosa, lymphoma, sporotrichosis and antiphospholipid syndrome.
* Classical systemic therapy (including but not limited to: corticosteroids, methotrexate, mycophenolate mofetil, azathioprine, tacrolimus, dapsone, cyclophosphamide) affecting pyoderma gangrenosum less than 14 days prior to enrollment.
* Therapy with other biologics (TNF antagonists, intravenous immunoglobulins) less than 3 months or 5 half-lives prior to enrollment, whichever is longer.
* Any other investigational drugs, other than investigational biologic treatment, within 30 days (or 3 months for investigational monoclonal antibodies) or 5 half-lives prior to the baseline visit, whichever is longer. Washout period may be longer according to local requirements.
* Topical therapy affecting pyoderma gangrenosum for a period of 14 days prior to enrollment.
* Having a history of recurring bacterial, viral, fungal, atypical mycobacterial infection, especially active or latent granulomatous infections (incl. tuberculosis, histoplasmosis) or currently undergoing treatment for tuberculosis.
* A positive quantiferon test indicating possible latent tuberculosis infection.
* An abnormal chest x-ray indicating a possible infection or malignoma for a period of 3 months prior to enrollment.
* Known Human Immunodeficiency Virus (HIV)-, Hepatitis B (HBV)-, or Hepatitis C (HCV)-infection.
* Having a severe medical condition that, in the judgment of the investigator, would jeopardize in any way the subject's safety following exposure to study drug.
* Pregnant or lactating women, patients (men or women) planning a pregnancy during the duration of the study, lack of safe contraception.

Safe contraception is defined as follows:

Double-barrier contraception such as oral, injectable, or implantable contraceptives, or intrauterine contraceptive devices together with condom use.

Both men and women must use safe contraception (double-barrier as defined above) during the duration of the study and until 6 months after the study.

Please note that female subjects who are surgically sterilized/hysterectomized or post-menopausal for longer than 2 years are not considered as being of child bearing potential.

* Having the presence or history of malignancy, including lymphoproliferative disorders. Subjects with a history of fully resolved basal or squamous cell skin cancer may be enrolled.
* Contraindications to monoclonal or polyclonal antibodies, e.g. known hypersensitivity or allergy to class of drugs or the investigational product.
* Known or suspected non-compliance, drug or alcohol abuse.
* Inability to follow the procedures of the study, e.g. due to language problems, psychological disorders, dementia or confusional state of the subject.
* Participation in another treatment study within the 30 days preceding and during the present study.
* Previous enrollment into the current study.
* Enrollment of the investigator, his/her family members, employees and other dependent persons.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2011-02; Primary Completion 2014-08 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Change of the Physician's global assessment (Grade 0-4) of the target lesion | Week 2, 4, 8, 16
  The primary response parameter change of the physician global assessment (PGA) 5-point scale at week 2, 4, 8, 16 as compared to week 0 :
  0= Total resolution of target ulcer with no signs of active PG
  1. Almost completely healed target ulcer with only minimal signs of active PG
  2. Evidence of target ulcer healing which involves at least 50% of ulcer/ulcer margin
  3. Evidence of target ulcer healing which involves less than 50% of ulcer/ulcer margin
  4. No evidence of target healing ulcer

SECONDARY OUTCOMES:
Change in surface area of the target lesion of pyoderma gangrenosum | Week 2, 4, 8, 16
  As secondary parameter, the change in surface area of the target lesion of pyoderma gangrenosum at week 2, 4, 8, 16 as compared to week 0 will be assessed by measuring the two-dimensional surface by tracing the border of the lesions on transparent foil as well as with Canfield photography.
Change in surface area of the non-target lesions | Week 2, 4, 8, 16
  As secondary parameter, the change in surface area of the non-target lesions of pyoderma gangrenosum at week 2, 4, 8, 16 as compared to week 0 will be assessed by measuring the two-dimensional surface by tracing the border of the lesions on transparent foil as well as with Canfield photography.

CONTACTS AND LOCATIONS:
Overall Officials: Lars French, Prof MD, Principal Investigator — University Hospital Zurich, Division of Dermatology
Locations (1):
- Department of Dermatology, University Hospital Zurich, Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: Yes
The data are in the Publication Kolios et al. British Journal of Dermatology, 2015